CLINICAL TRIAL: NCT04439630
Title: Evaluation of Potentially Bioactive Foods With Regard to Their Effects on Cardiometabolic Test Markers and Cognitive Variables
Brief Title: Effects of Nopal Fractions on Postprandial Glucose Regulation and Appetite Variables in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Protokoll 2018/8-b
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Glucose Tolerance; Appetite Sensations
Keywords: healthy subjects; diabetes prevention; obesity prevention

STUDY DESIGN:
Intervention Model Description: randomised crossover study in healthy young adults with normal BMI
Who Masked: Participant
Masking Description: Participants knew which test products that were included in the study, but not the consumption order
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- reference (Sham Comparator): Test product without the active components
  Interventions: Dietary Supplement: Test product without the active components
- Nopal fraction 1 (Experimental): Fraction one out of two possible
  Interventions: Dietary Supplement: Nopal fractions
- Nopal fraction 2 (Experimental): Fraction two out of two possible
  Interventions: Dietary Supplement: Nopal fractions

INTERVENTIONS:
Dietary Supplement: Nopal fractions — Nopal flour were divided in two fractions and mixed in two different test breads
  Arms: Nopal fraction 1; Nopal fraction 2
Dietary Supplement: Test product without the active components — Test product without the active components
  Arms: reference

SUMMARY:
Postprandial effects of Nopal fractions on glucose and appetite regulation will be investigated in healthy humans, in a randomised controlled crossover trial

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* non-smokers
* diet accordance with the Nordic Nutrition Recommendations
* BMI: 18.5-25 kg/m2

Exclusion Criteria:

* metabolic disorders
* food allergies
* no probiotics or other food /supplement which may interfere with the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
postprandial glucose tolerance | 0-180 min after start of the meal
  effects on postprandial glucose tolerance after intake of test products at breakfast. Measurements were performed at fasting (time = 0 min) and at 15, 30, 45, 60, 90, 120, 150 and 180 min.
postprandial insulin concentrations | 0-180 min
  effects on serum insulin concentrations after intake of test products at breakfast. Measurements were performed at fasting (time = 0 min) and at 15, 30, 45, 60, 90, 120, 150 and 180 min.

SECONDARY OUTCOMES:
subjective appetite variables | 0-180 min
  Subjective appetite variables (hunger, satiety, desire to eat) after intake of test products at breakfast, using a 100 mm Visual Analogue Scale (VAS) on a white paper. Except from a center mark in the center of the scale there was no other visible marks. Measurements were performed at fasting (time = 0 min) and at 15, 30, 45, 60, 90, 120, 150 and 180 min.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, assoc. prof., Principal Investigator — Lund University
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No